CLINICAL TRIAL: NCT00814229
Title: Randomised Dose Ranging Observer Blind Single Centre Study to Evaluate Safety and Immunogenicity of Adjuvanted and Non-adjuvanted Influenza H9 Influenza Vaccine in Humans
Brief Title: Safety and Immunogenicity of Influenza H9 Vaccine in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Crucell Holland BV (Industry); National Institute of Biological Standards and Control (Other Government); Public Health England (Other Government)
Responsible Party: Profressor Karl Nicholson, University of Leicester
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: UHL 08162; REC 6794
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Influenza
Keywords: influenza; H9N2; vaccine
MeSH Terms: conditions — Influenza, Human | interventions — aluminum sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (14):
- Vaccine 1 (Active Comparator): influenza H9N2 vaccine whole virus containing 1.5microg haemagglutinin by intramuscular injection
  Interventions: Biological: H9N2 whole virus vaccine, IM, 1.5microg
- vaccine 2 (Active Comparator): influenza H9N2 vaccine whole virus containing 5microg haemagglutinin by intramuscular injection
  Interventions: Biological: H9N2 whole virus vaccine, IM, 5microg
- Vaccine 3 (Active Comparator): influenza H9N2 vaccine whole virus containing 15microg haemagglutinin by intramuscular injection
  Interventions: Biological: H9N2 whole virus vaccine vaccine, IM, 15microg
- Vaccine 4 (Active Comparator): influenza H9N2 vaccine whole virus containing 45microg haemagglutinin by intramuscular injection
  Interventions: Biological: H9N2 whole virus vaccine, IM, 45microg
- Vaccine 5 (Active Comparator): influenza H9N2 vaccine whole virus adjuvanted with alum hydroxide containing 1.5microg haemagglutinin by intramuscular injection
  Interventions: Biological: H9N2 whole virus vaccine, alum, IM, 1.5microg
- Vaccine 6 (Active Comparator): influenza H9N2 vaccine whole virus adjuvanted with alum hydroxide containing 5microg haemagglutinin by intramuscular injection
  Interventions: Biological: H9N2 whole virus, alum, IM, 5microg
- Vaccine 7 (Active Comparator): influenza H9N2 vaccine whole virus adjuvanted with alum hydroxide containing 15microg haemagglutinin by intramuscular injection
  Interventions: Biological: H9N2 vaccine, whole virus, alum, IM, 15 microg
- Vaccine 8 (Active Comparator): influenza H9N2 vaccine whole virus adjuvanted with alum hydroxide containing 45microg haemagglutinin by intramuscular injection
  Interventions: Biological: H9N2 vaccine, whole virus, alum, IM, 45microg
- Vaccine 9 (Active Comparator): influenza H9N2 vaccine virosomal containing 1.5microg haemagglutinin by intramuscular injection
  Interventions: Biological: H9N2 virosome vaccine, IM, 1.5microg
- Vaccine 10 (Active Comparator): influenza H9N2 vaccine virosomal containing 5microg haemagglutinin by intramuscular injection
  Interventions: Biological: H9N2 virosomal vaccine, IM, 5microg
- Vaccine 11 (Active Comparator): influenza H9N2 vaccine virosomal containing 15microg haemagglutinin by intramuscular injection
  Interventions: Biological: H9N2 virosomal vaccine, IM, 15microg
- Vaccine 12 (Active Comparator): influenza H9N2 vaccine virosomal containing 45microg haemagglutinin by intramuscular injection
  Interventions: Biological: H9N2 virosomal vaccine, IM, 45microg
- Vaccine 13 (Active Comparator): influenza H9N2 vaccine whole virus containing 5microg haemagglutinin by intradermal injection
  Interventions: Biological: H9N2 whole virus vaccine, ID, 5microg
- Vaccine 14 (Active Comparator): influenza H9N2 vaccine whole virus containing 15microg haemagglutinin by intradermal injection
  Interventions: Biological: H9N2 whole virus vaccine, ID, 15microg

INTERVENTIONS:
Biological: H9N2 whole virus vaccine, IM, 1.5microg — influenza H9N2 vaccine whole virus containing 1.5microg haemagglutinin by intramuscular injection
  Arms: Vaccine 1
Biological: H9N2 whole virus vaccine, IM, 5microg — influenza H9N2 vaccine whole virus containing 5microg haemagglutinin by intramuscular injection
  Arms: vaccine 2
Biological: H9N2 whole virus vaccine vaccine, IM, 15microg — influenza H9N2 vaccine whole virus containing 15microg haemagglutinin by intramuscular injection
  Arms: Vaccine 3
Biological: H9N2 whole virus vaccine, IM, 45microg — influenza H9N2 vaccine whole virus containing 45microg haemagglutinin by intramuscular injection
  Arms: Vaccine 4
Biological: H9N2 whole virus vaccine, alum, IM, 1.5microg — influenza H9N2 vaccine whole virus adjuvanted with alum hydroxide containing 1.5microg haemagglutinin by intramuscular injection
  Arms: Vaccine 5
Biological: H9N2 whole virus, alum, IM, 5microg — influenza H9N2 vaccine whole virus adjuvanted with alum hydroxide containing 5microg haemagglutinin by intramuscular injection
  Arms: Vaccine 6
Biological: H9N2 vaccine, whole virus, alum, IM, 15 microg — influenza H9N2 vaccine whole virus adjuvanted with alum hydroxide containing 15microg haemagglutinin by intramuscular injection
  Arms: Vaccine 7
Biological: H9N2 vaccine, whole virus, alum, IM, 45microg — influenza H9N2 vaccine whole virus adjuvanted with alum hydroxide containing 45microg haemagglutinin by intramuscular injection
  Arms: Vaccine 8
Biological: H9N2 virosome vaccine, IM, 1.5microg — influenza H9N2 vaccine virosomal containing 1.5microg haemagglutinin by intramuscular injection
  Arms: Vaccine 9
Biological: H9N2 virosomal vaccine, IM, 5microg — influenza H9N2 vaccine virosome containing 5microg haemagglutinin by intramuscular injection
  Arms: Vaccine 10
Biological: H9N2 virosomal vaccine, IM, 15microg — influenza H9N2 vaccine virosome containing 15microg haemagglutinin by intramuscular injection
  Arms: Vaccine 11
Biological: H9N2 virosomal vaccine, IM, 45microg — influenza H9N2 vaccine virosome containing 45microg haemagglutinin by intramuscular injection
  Arms: Vaccine 12
Biological: H9N2 whole virus vaccine, ID, 5microg — influenza H9N2 vaccine whole virus containing 5microg haemagglutinin by intradermal injection
  Arms: Vaccine 13
Biological: H9N2 whole virus vaccine, ID, 15microg — influenza H9N2 vaccine whole virus containing 15microg haemagglutinin by intradermal injection
  Arms: Vaccine 14

SUMMARY:
H9N2 influenza circulates in animal and poultry and has caused delf limiting infections in children. Influenza H9N2 poses a pandemic threat to humans.

This study evaluates the safety and immunogenicity of adjuvanted and non-adjuvanted whole virus and virosomal H9N2 vaccines by the intramuscular route. We also assess intradermal route of administration to see if this has any advantages. The aim is to assess antibody responses before and after vaccination. The hypothesis is that lower doses of adjuvanted vaccine will induce similar antibody responses to non-adjuvanted vaccine

DETAILED DESCRIPTION:
A double-blind, single centre comparative study in which fourteen groups of 40 male and female adults >18 years of age will be randomly allocated to receive 1.7, 5, 15 or 45 µg quantities of whole virion (WV), Aluminium -adjuvanted WV(Al-WV), and virosomal (V) influenza A/Hong Kong/1073/99 (H9N2) vaccines by intramuscular injection into the deltoid muscle; or 5 or 15microg WV vaccine administered by intradermal injection. A second dose of the same vaccine containing the same quantity of antigen as in the first dose will be administered 21 days later. Subjects will be observed for local and systemic reactions for 30 minutes after each immunisation (day 0 and 21), and will be monitored for any reactions and other adverse events for 7 days after immunisation. Blood for immunogenicity studies will be obtained at day 0 (pre-immunisation), day-21 (+4 days), and at day-42 (i.e., 21 +4 days after the second immunization). Immunogenicity will be evaluated by haemagglutination inhibition, virus neutralization,, single radial haemolysis, neuraminidase inhibition and cellular mediated responses (in a subset of 5-10 subjects from each group).

ELIGIBILITY:
Inclusion Criteria:

* Mentally competent adults, who have signed an informed consent form after having received a detailed explanation of the study protocol.
* Male or female subjects over 18 years who are either healthy or have a stable medical condition.
* Able to understand and comply with all study procedures and to complete study diaries
* Individuals who can be contacted throughout the study and are available for all study visits
* Females should either be using secure contraceptive precautions including a) the oral contraceptive pill, b) condom/barrier contraception c) partner has had a vasectomy, d) be surgically sterilised, or e) post- (defined as at least two years since the last menstrual period)

Exclusion Criteria:

* Any clinically significant concurrent illness or unstable medical condition including: malignant tumours, autoimmune illnesses (including rheumatoid arthritis), acute or progressive renal or hepatic pathology, chronic obstructive pulmonary disease requiring oxygen therapy, and any active neurological disorder.
* Individuals with a history of anaphylaxis or serious reactions to vaccines; hypersensitivity to eggs, chicken protein, chicken feathers, influenzal viral protein, neomycin or polymixin, or products containing mercury.
* Persons with known immunosuppressive disease or who use systemic immunosuppressive drugs or other drugs listed in section 8 of the British National Formulary (BNF) or chloroquine, gold or penicillamine or other drugs listed in section 10.1.3 of the BNF to suppress a chronic disease process, or have received in the last 6 months radiotherapy or chemotherapy.
* Subjects who are at high risk of developing illnesses of the immune system.
* Individuals who are taking immunostimulant therapy or interferon
* Individuals who have received blood products or immunoglobulins parenterally during the preceding three months.
* Women should not be pregnant or lactating.
* Women who refuse to use a reliable contraceptive method throughout the study
* Known or suspected drug abuse.
* Individuals who have received another vaccine or experimental (investigational) drug in the preceding 4 weeks.
* Individuals who have previously received H9N2 vaccine
* Unable to lead an independent life either physically or mentally
* Regularly drink more than 40 units of alcohol weekly
* Individuals who have had acute respiratory pathology or infections requiring systemic antibiotic or antiviral therapy during the preceding 7 days (chronic antibiotic therapy for prevention of urinary tract infections is acceptable).
* Individuals who had a temperature over 38 degrees C in the preceding 3 days.
* Individuals who, in the opinion of the investigator, have conditions that might complicate interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Geometric mean antibody titres of antibody to influenza H9 by HI and neutralising antibody assays | Pre vaccination, 21 days and 42 days

SECONDARY OUTCOMES:
Local and systemic reactogenicity of influenza H9 vaccine | within 7 days of vaccination
seroprotective antibody titres to influenza H9 by HI and neutralising antibody | pre vacciantion, 21 and 42 days post-vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Karl G Nicholson, FRCP, MD, Principal Investigator — University of Leicester
Locations (1):
- University Hospitals Leicester, Leicester, Leicestershire, United Kingdom